CLINICAL TRIAL: NCT02126384
Title: Analysis of the Response of Healthy Adults to a 23-valent Pneumococcal Polysaccharide Vaccine to Identify the B Cell Subsets Responsible for the Production of IgM, IgG2 and IgA Anti-pneumococcal Capsular Polysaccharides
Brief Title: Identifocation the B Cell Subsets Responsible for Anti-pneumococcal Response
Acronym: PNEUMOVACB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INSERM-C12-10; 2013-000850-23 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-30 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2021-08

CONDITIONS: Pneumococcal Diseases
Keywords: Immunology; human; B-lymphocytes subsets; Antibody-Producing Cells; 23 valent pneumococcal capsular polysaccharide vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pneumovax (Experimental): Single arm, open label pneumovax vaccination of healthy subjects
  Interventions: Drug: pneumovax vaccination

INTERVENTIONS:
Drug: pneumovax vaccination — vaccination
  Other Names: pneumovax

SUMMARY:
The purpose of this study is to determine which B lymphocytes subsets are responsible for the production of IgM, IgG2 and IgA anti-pneumococcal capsular polysaccharides after vaccination with a 23-valent pneumococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
The aim of this study is to identify which specific B cell subset(s) is/are responsible for the production of protective IgM, IgG2 and IgA anti-pneumococcal capsular polysaccharides (capPS) in response to immunization of healthy individuals with the Pneumovax, a prototypical T-independent type 2 vaccine. In other words, from which B cells are IgM, G2 and A-secreting plasma cells derived? To address this question, it will be taken advantage of the unique Ig heavy chain VDJ signature expressed by each B cell clone and the strategy will rely on the search of clonal filiations between plasmablasts (PB)/plasma cells (PC) and different B cell subpopulations. Therefore, healthy individuals will be vaccinated with Pneumovax, and blood samples will be collected at day 0, 7, 14, 28 and 56. Starting from these blood samples, different B cells subsets (in particular IgM+IgD+CD27+ and switched memory IgM-IgD-CD27+ B cells) and the PB/PC peaking at day 7 after vaccination will be isolated by cell sorting. CapPS-secreting PB cannot be specifically isolated, but the investigators assume that they will represent the majority of the isolated PB/PC at the peak of the response. Thus, day 7-PB/PC will be sorted both in bulk or as single cells in 96-well PCR plates. RNA will be extracted from bulk sorted PB/PC, and VDJ-µ, -alpha and -gamma Ig transcripts will be amplified by RT-PCR and analyzed by the H-CDR spectratyping method in order to identify the sequence of dominant VDJ signatures that most probably correspond to anti-capPS-secreting cells. In parallel, for each PB/PC single cell, Ig heavy and corresponding Ig light chain gene transcripts will be amplified by nested RT-PCR, sequenced, and provided that the heavy chain contains a dominant VDJ signature, they will be cloned into eukaryotic expression vectors to produce monoclonal human Abs. The recombinant antibodies will then be tested for reactivity against capPS from the vaccine by ELISA. When VDJ signatures of capPS will be validated, with this powerful molecular tool, the investigators will look for the presence of these signatures through VDJ-specific PCR on cDNA prepared from the different B cell subsets.

ELIGIBILITY:
Inclusion Criteria:

* male
* aged 18 to 40 y

Exclusion Criteria:

* no documented primary immunodeficiency
* no splenectomy
* no functional/congenital asplenia,
* no pneumococcal infections within the last 5 years before enrolment into the research protocol
* no vaccinations with the 23-valent pneumococcal polysaccharide vaccine or the 7- or 13-valent conjugate-polysaccharide vaccines within the last 5 years before enrolment into the research protocol
* no other vaccination within 1 month before enrolment into the research protocol
* fever, current antibiotic treatment
* any chronic or inflammatory disease
* any immunosuppressive treatment
* hyper-responsiveness to one component of the Pneumovax vaccine

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Identification of the precursor of B lymphocytes | day 7
  On vitro measure of blood mononuclear cell populations by cell sorting at day 7 to identify the clonal progeny of the secreting B lymphocyte precursor

SECONDARY OUTCOMES:
measure of serum anti-capsular polysaccharide antibody titers | day 0, day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sandra WELLER, PhD, Study Director — Institut National de la santé et de la recherché Médicale (INSERM)
Locations (1):
- Centre d'Investigation Clinique, hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Weller S, Sterlin D, Fadeev T, Coignard E, Verge de Los Aires A, Goetz C, Fritzen R, Bahuaud M, Batteux F, Gorochov G, Weill JC, Reynaud CA. T-independent responses to polysaccharides in humans mobilize marginal zone B cells prediversified against gut bacterial antigens. Sci Immunol. 2023 Jan 27;8(79):eade1413. doi: 10.1126/sciimmunol.ade1413. Epub 2023 Jan 27. PMID 36706172